CLINICAL TRIAL: NCT00002697
Title: HIGH DOSE CHEMORADIOTHERAPY WITH PERIPHERAL BLOOD PROGENITOR CELL TRANSPLANTATION FOR PATIENTS WITH PRIMARY REFRACTORY, RELAPSED AND POOR PROGNOSIS NON-HODGKIN'S LYMPHOMA
Brief Title: Combination Chemotherapy Plus Radiation Therapy Followed by Peripheral Stem Cell Transplantation in Treating Patients With Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Masking: None | Purpose: Treatment
Other Study IDs: 95-072; CDR0000064483 (Registry Identifier: PDQ (Physician Data Query)); NCI-V95-0784
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Filgrastim; sargramostim; Carboplatin; Etoposide; Ifosfamide; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Biological: sargramostim
Drug: carboplatin
Drug: etoposide
Drug: ifosfamide
Procedure: autologous bone marrow transplantation
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with radiation therapy and peripheral stem cell transplantation may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of high-dose combination chemotherapy plus radiation therapy followed by peripheral stem cell transplantation in patients with refractory or recurrent non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of mobilization using filgrastim (G-CSF) with or without standard-dose ifosfamide, carboplatin, and etoposide (ICE), conditioning using ifosfamide and etoposide plus total body irradiation or high-dose ICE, and autologous peripheral blood stem cell (PBSC) transplantation as salvage therapy in patients with refractory, recurrent, or poor prognosis non-Hodgkin's lymphoma.
* Determine the efficacy of reinduction comprising ICE followed by autologous PBSC transplantation in these patients.
* Determine the ability of standard-dose ICE combined with hematopoietic growth factors to mobilize PBSC in these patients.
* Determine the contamination of PBSC by lymphoma cells in patients treated with this mobilization regimen.
* Determine the quality of life of patients treated with this regimen.

OUTLINE: Patients are stratified according to disease status (relapsed vs refractory), lymphoma grade (low vs intermediate vs high), number of extranodal sites, serum lactic dehydrogenase, performance status, age, and volume of disease.

* Mobilization/harvest: Patients in first or greater complete remission (CR) are treated on regimen A, whereas patients with recurrent or refractory disease are treated on regimen B.

  * Regimen A: Patients with poor prognosis intermediate-grade lymphoma (IGL) in first CR or IGL or low-grade lymphoma (LGL) in second or greater CR receive mobilization with filgrastim (G-CSF) subcutaneously (SC) daily on days 1-7. Autologous peripheral blood stem cells (PBSC) are harvested and selected for CD34+ cells on days 5 and 6 (and day 7 if needed).
  * Regimen B: Patients who are currently on the MSKCC standard dose salvage therapy protocol with ifosfamide, carboplatin, and etoposide (ICE) for recurrent or refractory IGL receive additional mobilization with G-CSF after completion of the last course of ICE. Patients with recurrent or refractory IGL, immunoblastic lymphoma, or LGL who have not previously received ifosfamide and are not currently on the MSKCC standard dose salvage protocol with ICE receive ifosfamide IV and carboplatin on day 2 and etoposide IV on days 1-3 (standard-dose ICE) followed by G-CSF SC. When blood counts recover, autologous PBSC are harvested and selected for CD34+ cells.
  * Regimens A and B: If additional hematopoietic growth factors (HGFs) become available, they may be administered concurrently with G-CSF. If inadequate CD34+ cells are collected, then autologous bone marrow is harvested.
* Conditioning: Patients who are under age 60 and have not received dose-limiting radiotherapy are treated on regimen C. Patients who are age 60 and over and patients who are under age 60 and have received dose-limiting radiotherapy are treated on regimen D.

  * Regimen C: Patients undergo hyperfractionated total body irradiation twice a day on days -10 to -7 and ifosfamide IV over 1 hour followed by etoposide IV over 23 hours on days -6 to -2.
  * Regimen D: Patients receive ifosfamide IV over 1 hour, followed by etoposide IV over 11 hours, followed by carboplatin IV over 1 hour, followed by etoposide IV over 11 hours on days -7 to -3 (high-dose ICE).
  * Regimens C and D: Patients with residual or relapsed disease may undergo boost radiotherapy twice a day, 5 days a week, for 1-2 weeks before conditioning or after transplantation.
* Transplantation: PBSC or bone marrow is reinfused on day 0. Patients receive G-CSF SC every 12 hours beginning on day 1 and continuing until blood counts recover. If additional HGFs become available, they may be administered concurrently with G-CSF.

Quality of life is assessed at baseline and then at 6, 12, and 24 months after transplantation.

Patients are followed at 1 and 3 months, every 3 months through year 2, every 4 months through year 5, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 80 patients (20 for regimen A and 60 for regimen B) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following diagnoses:

  * Histologically proven recurrent non-Hodgkin's lymphoma

    * Previously in complete remission (CR)
  * Refractory or recurrent intermediate-grade lymphoma (IGL) or high-grade immunoblastic lymphoma (IBL) meeting 1 of the following conditions:

    * In partial remission (PR) or CR to and currently enrolled on the MSKCC standard dose salvage regimen with ifosfamide, carboplatin, and etoposide (ICE)
    * In PR or CR after 1-2 other salvage chemotherapy regimens (e.g., 3 courses of dexamethasone, high-dose cytarabine, and cisplatin (DHAP); 2 courses of cyclophosphamide, mechlorethamine, vincristine, procarbazine, and prednisone (C-MOPP))

      * No prior ifosfamide
  * Low-grade lymphoma

    * In second or greater remission or chemosensitive relapse
    * No HLA identical sibling donor available
  * IGL or IBL

    * In first CR
    * Poor prognosis, defined by age-adjusted international index of 3 or 4 based on lactic dehydrogenase, number of extranodal sites, stage, and performance status
* Adequate bone marrow cellularity
* No lymphoblastic or small noncleaved cell lymphoma
* Ineligible for total body irradiation (TBI) phase of study if prior radiotherapy dose precludes the use of TBI NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma.However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age:

* Physiologic 18 to 65

Performance status:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 2.0 mg/dL (if no history of Gilbert's disease)
* No chronic active or persistent hepatitis
* Hepatitis B positivity allowed provided that the following conditions are met:

  * Bilirubin same as above*
  * SGPT no greater than 500 IU/L*
  * Alkaline phosphatase no greater than 2 times normal* NOTE: * In the absence of liver involvement by lymphoma

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min
* No history of chronic renal insufficiency

Cardiovascular:

* LVEF at least 50% by echocardiogram or MUGA scan
* No myocardial infarction within the past 6 months
* No unstable angina
* No arrhythmia other than chronic atrial fibrillation

Pulmonary:

* DLCO at least 50% predicted (corrected for hemoglobin and alveolar ventilation)

Other:

* HIV negative
* No uncontrolled infection
* No other malignancy within the past 5 years except curatively treated basal cell skin cancer or carcinoma in situ of the cervix
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics

Surgery

* Not specified

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1995-09; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Moskowitz, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States